CLINICAL TRIAL: NCT00725998
Title: Longitudinal Study Of The Evoked Compound Action Potential Measured In Children Cochlear Implant Users
Acronym: ECAP
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Other Study IDs: CEP 039/2004
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2008-07

CONDITIONS: Cochlear Nerve Disease
Keywords: Cochlear Implantation.; Cochlear nerve.; Child.; study; ECAP; During; First year
MeSH Terms: conditions — Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- 1: The ECAP characteristics have been analyzed in 13 children implanted younger than three years old.
  Series Study Results:
  During the first year of CI use there was a significant statistical growth for the amplitude of N1 peak, in basal electrodes, between the second and third returns. There were not any significant differences obtained for N1 peak, latency, slope, neither for p-NRT nor recovery time, among the returns.

SUMMARY:
Introduction: In Cochlear Implant (CI) users, the recording of the electrically evoked compound action potential (ECAP) of the auditory nerve represents an option to assess changes in auditory nerve responses and the interaction between the electrode and the neural tissue over time.

Aim: To study ECAP in children during the first year of CI use.

Material and methods: The ECAP characteristics have been analyzed in 13 children implanted younger than three years old. SERIES STUDY.

Descriptors:

Cochlear Implantation,cochlear nerve,child.

ELIGIBILITY:
This study selected only children implanted younger than three years old and followed them during their first year of CI use.

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The ECAP characteristics have been analyzed in 13 children implanted younger than three years old.
Sampling Method: Non-Probability Sample
Dates: Start 2005-01; Primary Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de São Paulo, Bauru, São Paulo, Brazil